CLINICAL TRIAL: NCT01211379
Title: The FLU-FOBT Program: Translation of an Evidence-Based Colorectal Cancer Screening Program to Primary Care Settings Where Disparities Persist
Brief Title: The FLU-FOBT Program in Primary Care Settings Where Disparities Persist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Department of Public Health (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Michael B. Potter, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1R18DP001566-01 (NIH)
Record Dates: First submitted 2010-09-25; First posted 2010-09-29 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-09

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer screening; primary care; health disparities
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FLU-Only Arm (No Intervention): In this arm, primary care patients who got flu shots were only provided with FOBT if the doctor decided to order it.
- FLU-FOBT Arm (Experimental): In this arm, patients who came in for primary care got a flu shot and were assessed by nurses for eligibility for colorectal cancer screening. Eligible patients were provided with home FOBT.
  Interventions: Behavioral: FLU-FOBT Program

INTERVENTIONS:
Behavioral: FLU-FOBT Program — Primary care patients who came in for flu shots were assessed by nurses for colorectal cancer screening eligibility and offered FOBT if due.
  Arms: FLU-FOBT Arm

SUMMARY:
The investigators overall goals are to adapt, implement, evaluate, and disseminate the FLU-FOBT Program as an integrated nurse-run, primary care-based intervention that can reduce colorectal cancer screening disparities in resource-poor clinical settings. In this program, fecal occult blood tests (FOBT) are provided with influenza vaccinations (FLU) to eligible patients between the ages of 50 and 75 during FLU season. The investigators hypothesis is that the FLU-FOBT Program can be adapted for primary care settings and lead to higher rates of colorectal cancer screening (CRCS).

DETAILED DESCRIPTION:
AIM 1 (Year 1): To adapt and pilot test the FLU-FOBT Program as a nurse-run intervention during primary care visits at San Francisco's Chinatown Public Health Center. The FLU-FOBT Program will be designed in such a way as to trigger the offering of fecal occult blood testing (FOBT) to eligible patients whenever an influenza vaccination (FLU) is provided. Specific components of the FLU-FOBT Program will be developed through a process of active collaboration with health center staff. The FLU-FOBT Program will be implemented in the fall of 2008-9 and evaluated with a combination of process measures in Year 1 of the study. This formative work will be used to finalize the FLU-FOBT Program for further study of its efficacy and robustness in other affiliated San Francisco public health centers.

AIM 2 (Year 2 and 3): To test the efficacy of the FLU-FOBT Program in improving colorectal cancer screening rates in a time-randomized, controlled trial involving other public health centers in the San Francisco Community Health Network that serve ethnically diverse, economically disadvantaged patients. During the 2009-10 influenza vaccination season, the FLU-FOBT Program will be tested in a randomized trial within 6 public health centers in San Francisco. On half of randomly selected dates at each of these clinics, a nurse will follow a protocol that directs them to offer FOBT to eligible patients whenever they are offered an influenza vaccine (intervention), and on the other dates nurses will be directed to offer just influenza vaccine alone (control). The primary efficacy outcome will be the proportion of intervention subjects between the ages of 50 and 80 and are initially due for CRCS who become up to date 3 months after the intervention is completed, as compared with similar subjects in the control group.

AIM 3 (Years 2 and 3): To evaluate the robustness of the FLU-FOBT Program as implemented within these 6 clinics. In the 2009-10 influenza vaccination season, we will also test the robustness of the FLU-FOBT Program as implemented at the 6 sites that participate in the time-randomized trial. Robustness will be measured according to the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation, and Maintenance) described by Glasgow and others [2]. Reach will be measured as the proportion of the target population that is offered screening, and Effectiveness will be measured as the proportion of the target population that gets screened with the intervention. Adoption will be measured as the proportion of invited influenza vaccination clinic sites and clinic staff members that participate; Implementation will be assessed according to the fidelity with which participating sites and clinic staff follow the key elements of FLU-FOBT Program protocol and how they adapt the protocol to accommodate local needs and constraints. Maintenance will be assessed by determining the number of intervention sites that continue the FLU-FOBT Program in the year after the intervention has been completed, and the overall success of the program where it is continued.

AIM 4 (Year 3): To develop a FLU-FOBT Program Toolkit that can be adopted locally and disseminated to other public health clinics that rely on annual FOBT as a primary strategy for average risk colorectal cancer screening. Study results from all participating health centers will be used to develop an evidence-based FLU-FOBT Toolkit that can be distributed and serve as a practical guide for clinical decision makers who wish to adapt and replicate this intervention within clinics that serve diverse communities that experience disparities in colorectal cancer screening. The Toolkit will include both key elements that must be preserved in order for the FLU-FOBT Program to be successful, as well as examples of enhancements successfully implemented in different clinics

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be primary care patients one of 6 participating clinics
2. Participants must be aged 50-75
3. Participants must have received a flu shot during a primary care visit on any date during the 2009-10 flu shot season (beginning September 28, 2009 and ending at the end of January, 2010).

Exclusion Criteria: None

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1372 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change in Colorectal Cancer Screening Rate | March 30, 2010
  Change in colorectal cancer screening rates (defined as being up to date with FOBT in the last 12 months, up to date with flexible sigmoidoscopy within the last 5 years, or up to date with colonoscopy in the last 10 years) by March 30, 2010, 6 months after the beginning of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Potter, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Department of Public Health, San Francisco, California, United States

REFERENCES:
- [Derived] Potter MB, Walsh JM, Yu TM, Gildengorin G, Green LW, McPhee SJ. The effectiveness of the FLU-FOBT program in primary care a randomized trial. Am J Prev Med. 2011 Jul;41(1):9-16. doi: 10.1016/j.amepre.2011.03.011. PMID 21665058